CLINICAL TRIAL: NCT01212471
Title: A Dose Ranging Study to Evaluate Safety and Efficacy of Bromfenac Ophthalmic Solution in Dry Eye Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S00007
Record Dates: First submitted 2010-09-28; First posted 2010-09-30 (Estimated); Results first posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Dry Eye Syndrome
Keywords: Sign and symptoms of dry eye disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bromfenac Ophthalmic Solution A (Experimental): Bromfenac ophthalmic solution A
  Interventions: Drug: Bromfenac Ophthalmic Solution A
- Bromfenac Ophthalmic Solution B (Experimental): Bromfenac ophthalmic solution B
  Interventions: Drug: Bromfenac Ophthalmic Solution B
- Placebo Comparator (Placebo Comparator): Placebo Comparator
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Bromfenac Ophthalmic Solution A — sterile ophthalmic solution
  Arms: Bromfenac Ophthalmic Solution A
Drug: Bromfenac Ophthalmic Solution B — sterile ophthalmic solution
  Arms: Bromfenac Ophthalmic Solution B
Drug: Placebo Comparator — sterile ophthalmic solution
  Arms: Placebo Comparator

SUMMARY:
A dose ranging study to evaluate safety and efficacy of bromfenac ophthalmic solution in dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Be of either gender and any race 18 years or older

Exclusion Criteria:

* Have a local or systemic disease that could interfere with the assessment of safety or efficacy or that is likely to result in early discontinuation from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Actual)
Dates: Start 2010-09; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim McNamara, PharmD, Study Director — ISTA Pharmaceuticals, Inc.
Locations (1):
- ISTA Pharmaceuticals, Inc., Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bromfenac Ophthalmic Solution 0.06%: Bromfenac Ophthalmic Solution 0.06% twice a day
- Bromfenac Ophthalmic Solution 0.03%: Bromfenac Ophthalmic Solution 0.03% twice a day
Period: Overall Study
Arm/Group | Bromfenac Ophthalmic Solution 0.06% | Bromfenac Ophthalmic Solution 0.03% | Placebo Comparator
Started | 141 | 140 | 139
Completed | 139 | 137 | 132
Not Completed | 2 | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bromfenac Ophthalmic Solution 0.06% | Bromfenac Ophthalmic Solution 0.03% | Placebo Comparator | Total
Number analyzed (Participants) | 141 | 140 | 139 | 420
Age, Continuous [Mean (Full Range); unit: years] | 61.0 [19 to 89] | 61.6 [21 to 89] | 61.0 [26 to 84] | 61.2 [19 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 112 | 112 | 333
  Male | 32 | 28 | 27 | 87

OUTCOME MEASURES:

1. Primary Outcome: Mean Ocular Surface Disease Index (OSDI) Total Score
Description: The Ocular Surface Disease Index (OSDI) is a 12 item questionnaire. Each question about discomfort/limitations is scored from 0 to 4, with 0 being 'None of the Time' and 4 being 'All of the Time'. The minimum total score is 0 and the maximum total score is 48, with higher scores indicating worse outcomes.
Time Frame: 42 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bromfenac Ophthalmic Solution 0.06% | Bromfenac Ophthalmic Solution 0.03% | Placebo Comparator
Number analyzed (Participants) | 141 | 140 | 139
score on a scale | 35.0 (22.23) | 40.3 (25.22) | 36.9 (23.24)

ADVERSE EVENTS:
Time Frame: 10 days
Arm/Group | Bromfenac Ophthalmic Solution 0.06% | Bromfenac Ophthalmic Solution 0.03% | Placebo Comparator
All-Cause Mortality (participants affected / at risk) | 0/141 | 0/140 | 0/139
Serious Adverse Events (participants affected / at risk) | 2/141 | 3/140 | 1/139
Other Adverse Events (participants affected / at risk) | 9/141 | 8/140 | 7/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bromfenac Ophthalmic Solution 0.06% (N=141) | Bromfenac Ophthalmic Solution 0.03% (N=140) | Placebo Comparator (N=139)
Carotid artery disease (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular event (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis atrophic (Gastrointestinal disorders) | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Adverse drug reaction (General disorders) | 0 | 0 | 1
Chest discomfort (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Mental status change (Psychiatric disorders) | 1 | 0 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bromfenac Ophthalmic Solution 0.06% (N=141) | Bromfenac Ophthalmic Solution 0.03% (N=140) | Placebo Comparator (N=139)
Dry eye (Eye disorders) | 9 | 8 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.